CLINICAL TRIAL: NCT04153877
Title: The Effect of Kinesio-tape® on Pain and Vertical Jump Performance in Active Individuals With Patellar Tendinopathy
Status: Completed | Type: Observational
Sponsor: University of Hawaii (Other)
Responsible Party: Principal Investigator, Kaori Tamura, Associate Professor, University of Hawaii
Other Study IDs: CHS#23178
Record Dates: First submitted 2019-11-01; First posted 2019-11-06 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Patellar Tendinitis
MeSH Terms: interventions — Athletic Tape

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Kinesiotape — Kinesio-tape® is an elastic, hypoallergenic, cotton-fiber tape with acrylic heat-activated backing and is widely used within sports.

SUMMARY:
Background: Patellar tendinopathy is a common inflammatory condition in athletes who undergo large volumes of running and jumping. Kinesio-tape® (KT) is proposed to provide pain relief; however, its effect has not been examined on patellar tendinopathy. Objective: To examine the effects of KT on pain modulation for active individuals with patellar tendinopathy during functional activities. Methods: Thirteen symptomatic knees from seven college-aged females (6 bilateral; 1 unilateral) were included. Participants underwent three data collection sessions with KT, sham, and no tape (NT) in a randomized order. During the session, participants performed a maximum vertical jump, single-leg squats and isometric knee extension. The KT intervention was applied according to the KT manual and the sham utilized the same pattern without tension. Pain level was evaluated using the numeric pain scale before, during and after each activity. Function was assessed as maximum vertical jump height and maximum isometric strength.

ELIGIBILITY:
Inclusion Criteria:

* Anterior knee pain that increases with jumping and/or squatting
* Pain with palpation at the tibial tuberosity, the patellar tendon, and/or at the apex of the patella
* An insidious onset of this pain.
* Participate in physical activity at least 3 days a week

Exclusion Criteria:

* Injury from direct trauma to the anterior knee
* Medical history of surgery at the knee joint within the past 6 months
* Presence of any lower extremity injuries or non-orthopedic diseases
* Suspected or confirmed pregnancy.

Ages: 18 Years to 30 Years | Sex: Female
Age Groups: Adult
Study Population: College-aged physically active female with patellar tendinopathy
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-03-28 (Actual); Study Completion 2017-04-28 (Actual)

PRIMARY OUTCOMES:
Change in pain level from no tape condition | at 3 different time point, with kinesiotape, sham tape, and not tape conditions, which are separated by 3 to 7 days
  measured using the Numeric Pain Scale ranging from zero to ten, with zero representing no pain, five as moderate pain and ten being unbearable pain.
Change in maximum vertical jump height from no tape condition | at 3 different time point, with kinesiotape, sham tape, and not tape conditions, which are separated by 3 to 7 days
  measured using a Vertec measurement system in inches
Change in maximum isometric strength from no tape condition | at 3 different time point, with kinesiotape, sham tape, and not tape conditions, which are separated by 3 to 7 days
  measured using a MicroFet2 Hand Held Dynamometer in Newton metre

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tamura K, Resnick PB, Hamelin BP, Oba Y, Hetzler RK, Stickley CD. The effect of Kinesio-tape(R) on pain and vertical jump performance in active individuals with patellar tendinopathy. J Bodyw Mov Ther. 2020 Jul;24(3):9-14. doi: 10.1016/j.jbmt.2020.02.005. Epub 2020 Feb 22. PMID 32826014